CLINICAL TRIAL: NCT02269241
Title: A Pivotal, Multicenter, Non-Comparative Trial on the Contraceptive Efficacy, Safety, Tolerability and Pharmacokinetics of LF111 (Drospirenone 4.0 mg) During 13 Cycles
Brief Title: Safety, Efficacy, Tolerability and Pharmacokinetics of LF111 (Drospirenone 4.0 mg) During 13 Cycles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratories Leon Farma, S.A. (Industry)
Collaborators: Chemo France (Industry)
Responsible Party: Sponsor
Organization: Insud Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF111/303
Record Dates: First submitted 2014-10-06; First posted 2014-10-21 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2017-10

CONDITIONS: Contraception
Keywords: contraception; hormonal oral contraceptive agents; hormonal oral contraceptive; oral contraceptive; drospirenone; LF111; birth control
MeSH Terms: interventions — drospirenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LF111 (drospirenone) (Experimental): single treatment arm receives LF111
  Interventions: Drug: LF111 (drospirenone)

INTERVENTIONS:
Drug: LF111 (drospirenone) — One LF111 tablet once per day for 24 days followed by 4 placebo tablets for 4 days equals one cycle.
  Other Names: CF111

SUMMARY:
To demonstrate the contraceptive efficacy of LF111 . To demonstrate the safety and tolerability of LF111 and assessment of pharmacokinetics of LF111.

DETAILED DESCRIPTION:
This trial is a prospective, multicenter, open-label, non-controlled trial in female subjects, including adolescents between the ages of 15+(inclusive) who present to the clinic seeking contraception, who are postmenarcheal and premenopausal.

At screening, informed consent will be obtained and the screening procedures will be performed. After confirmation of the subject's eligibility, the subject will be provided with the investigational product and trained in the use of an electronic diary. Afterwards, the subjects will attend visit the clinical site on Day 20±2 of the 1st, 3rd, 6th and 9th cycles and on Day 29+2 of the 13th cycle. The last clinical site visit will occur 10-14 days after the 13th cycle visit.

The trial will include women who have never used hormonal contraceptives before consent (naïve users), women who have not used hormonal contraceptives in the past three months before consent or who have used hormonal contraceptives in the past but have a contraceptive-free time of less than three months before consent (previous users) as well as women directly switching from another hormonal method (switchers). Women who have used hormonal contraceptives in the past but have a contraceptive-free time of less than three months before consent are allowed to be included into the trial if they had at least one complete menstrual cycle before enrollment.

A population pharmacokinetic (PK) analysis planned in the whole subject population, will obtain sparse blood samples to determine plasma concentrations. In total, four blood samples will be collected: two samples each will be collected during the 1st cycle and during the 6th cycle of treatment.

Adverse events and safety information will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Sexually active, postmenarcheal and premenopausal female subjects at risk of pregnancy including breastfeeding women with no upper age limit.
2. Female subjects at risk of pregnancy, between the ages of 15 and 17 (inclusive) provided that

   * Applicable national, state and local laws allow subjects in this age group to consent/assent to receive contraceptive services, and
   * All applicable laws and regulations regarding the informed consent/assent of the subjects to participate in clinical trials are observed.
3. Regular cycles during the last six months before consent/assent when not using hormonal contraception.
4. At least three complete menstrual cycles after delivery (only applicable for women who were pregnant within the last six months and for non-breastfeeding women). Breastfeeding women can be included six weeks after delivery irrespective of menstrual cycles post-delivery.
5. At screening, maximum systolic blood pressure (median value of three values) ≤ 159 mm Hg and diastolic blood pressure (median value of three values) ≤ 99 mm Hg.
6. Be able and willing to provide written informed consent or assent if the subject is adolescent, prior to undergoing any trial-related procedure.
7. Willing to use trial contraception for thirteen 28-day cycles.
8. Be willing to have intercourse each cycle of trial without the need to use back-up contraceptive.
9. Be willing to state that, to her best knowledge, her male sexual partner(s):

   * Has not had a vasectomy or been previously diagnosed as infertile.
   * Has not been previously diagnosed or suspected of human immunodeficiency virus (HIV) unless he has subsequently had a negative HIV test.
   * Has not been known to have engaged in homosexual intercourse in the past five years unless he has had negative HIV test results since then.
   * Has not shared injection drug needles in the past unless he has had a negative HIV test at least six weeks since last use.
10. Agree not to participate in any other clinical trials during the course of this trial.

Exclusion Criteria:

1. Pregnant.
2. Subject is known to or suspected of not being able to comply with the trial protocol, the use of the trial medication or the use of the trial diary.
3. History of infertility.
4. Abnormal finding on pelvic, breast or ultrasound examination that in the investigator's opinion contraindicates participation in the trial.
5. Unexplained amenorrhea.
6. Known polycystic ovary syndrome.
7. Women ≥21 years of age with a Papanicolaou (pap) smear reading LGSIL or higher at screening (or six months prior to screening date). Human papilloma virus (HPV) testing in subjects with atypical squamous cells of undetermined significance (ASC-US) can be used as an adjunctive test.

   * Subjects with ASC-US can be included if they are negative for high-risk HPV strains.
   * Subjects <21 years of age do not require a pap smear.
8. Known contraindication or hypersensitivity to ingredients or excipients of the IMP (Investigational Medicinal Product), including:

   1. Renal insufficiency
   2. Hepatic dysfunction
   3. Adrenal insufficiency
   4. Current or history of venous thrombophlebitis or thromboembolic disorders (venous thromboembolism, which includes deep vein thrombosis and pulmonary embolism)
   5. Current or history of cerebral-vascular or coronary-artery disease
   6. Valvular heart disease with thrombogenic complications
   7. Diabetes with vascular involvement
   8. Headaches with focal neurological symptoms
   9. Major surgery with prolonged immobilization
   10. Known or suspected carcinoma of the breast
   11. Known or suspected sex-steroid sensitive malignancies
   12. Undiagnosed abnormal genital bleeding
   13. Cholestatic jaundice of pregnancy or jaundice with prior hormonal contraceptive use
   14. Liver tumor (benign or malignant) or active clinically significant liver disease.
9. Uncontrolled thyroid disorder (i.e., on stable dose of thyroid replacement for less than two months).
10. Uncontrolled concomitant diseases (i.e., not on a stable treatment dose for at least two months).
11. Evidence or history of alcohol, medication or drug abuse (within the last 12 months prior to consent/assent).
12. Known inherited or acquired predisposition to venous thromboembolism or arterial thromboembolism (e.g., factor V Leiden, Prothrombin mutation, Antiphospholipid antibodies) or bruising within the last 12 months prior to consent/assent.
13. Known or suspected HIV and/or hepatitis infection at screening.
14. Received a dose of depot medroxyprogesterone acetate (DMPA or Depo-Provera®) during the 10 months prior to consent/assent, or received any combined injectable contraceptive (e.g., Cyclofem®) during the six months prior to consent/assent, or no spontaneous menses since last injection.
15. Long-term treatment (longer than seven consecutive days within a month prior to V1b) of any medication that might interfere with the efficacy of hormonal contraceptives.

    Prohibited medication include:
    1. Anticonvulsants (e.g. phenytoin, carbamazepine, oxcarbazepine, topiramate, felbamate, primidone)
    2. Barbiturates
    3. Rifampin
    4. Bosentan
    5. Griseofulvin
    6. St. John's wort (hypericum perforatum)
16. Administration of human chorionic gonadotropin (hCG) or intake of co-medication containing hCG within a month prior to V1b).
17. Progestin-releasing intra-uterine device (IUD) or contraceptive implant received or in place within the last two months prior to consent/assent.
18. Planned regular concomitant use of barrier contraceptive methods, spermicides, IUDs or other contraceptive measures (excepting occasional use for safety reasons, e.g., to reduce risk of infection).
19. Evidence or history of clinically significant psychiatric illness or suicide risk.
20. Participation in another trial of an investigational drug or device parallel to the current trial or less than 90 days before consent/assent, or previous participation in the current trial and dispensed trial medication.
21. Subject is a member of the investigator's or Sponsor's staff or a relative or family member thereof.
22. Any condition that, in the opinion of the investigator, may jeopardize protocol compliance or the scientific integrity of the trial.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1552 (Actual)
Dates: Start 2014-10-09 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Colli, MD, Study Director — Exeltis
Locations (37):
- United States (37):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - WCCT Global, Costa Mesa, California
  - Women's Health Care Research Corp., San Diego, California
  - Downtown Women's Health Care, Denver, Colorado
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Altus Research, Lake Worth, Florida
  - Miami Research Associates, Miami, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Meridien Research - St. Petersburg, St. Petersburg, Florida
  - Meridien Research - Tampa, Tampa, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Fellows Research Alliance, Inc., Savannah, Georgia
  - Rosemark WomenCare Specialists, Idaho Falls, Idaho
  - Bluegrass Clinical Research, Inc, Louisville, Kentucky
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Beyer Research, Kalamazoo, Michigan
  - Lawrence OBGYN Clinical Research, LLC, Lawrenceville, New Jersey
  - The Center for Women's Health & Wellness, LLC, Plainsboro, New Jersey
  - Southwest Clinical Research, Albuquerque, New Mexico
  - NYU School of Medicine, New York, New York
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Columbus Obstetricians-Gynecology, Inc./Radiant Research, Inc., Columbus, Ohio
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - Clinical Research Of Philadelphia, Philadelphia, Pennsylvania
  - Fellows Research Alliance, Inc., Bluffton, South Carolina
  - Advanced Research Associates, Corpus Christi, Texas
  - Practice Research Organization, Dallas, Texas
  - TMC Life Research, Inc., Houston, Texas
  - Physicians' Research Options, Draper, Utah
  - Physicians' Research Options, Pleasant Grove, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Seattle Women's Health, Research, Gynecology, Seattle, Washington

REFERENCES:
- [Derived] Palacios S, Colli E, Regidor PA. Efficacy and cardiovascular safety of the new estrogen-free contraceptive pill containing 4 mg drospirenone alone in a 24/4 regime. BMC Womens Health. 2020 Oct 2;20(1):218. doi: 10.1186/s12905-020-01080-9. PMID 33008401

RESULTS

PARTICIPANT FLOW:
Groups:
- Drospirenone 4 mg: Single treatment arm receives LF111 film-coated tablets (24 white tablets containing 4.0 mg drospirenone, 4 green placebo tablets), oral administration once daily.
Period: Overall Study
Arm/Group | Drospirenone 4 mg
Started | 1552
Completed | 352
Not Completed | 1200
Not completed — Lost to Follow-up | 269
Not completed — Withdrawal by Subject | 155
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 7
Not completed — Pregnancy | 15
Not completed — Wish for pregnancy | 5
Not completed — Development of an exclusion criteria | 16
Not completed — Adverse Event | 113
Not completed — At the specific request of the sponsor | 20
Not completed — Several reasons not classified | 53
Not completed — Screening failures | 546

BASELINE CHARACTERISTICS:
Population: 1552 patients enrolled, 546 patients screening failures, 1006 patients analyzed, 352 patients completed
Groups:
- LF111 (Drospirenone 4mg): Single treatment arm receives LF111 film-coated tablets (24 white tablets containing 4.0 mg drospirenone, 4 green placebo tablets), oral administration once daily.
Arm/Group | LF111 (Drospirenone 4mg)
Number analyzed (Participants) | 1006
Age, Customized [Number; unit: participants]
  <=35 years | 928
  >35 years | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1006
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 229
  Not Hispanic or Latino | 777
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 5
  Black or African American | 358
  White | 571
  More than one race | 0
  Unknown or Not Reported | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Pregnancies (Evaluable Cycles)
Description: Pearl index (PI) from Evaluable Cycles in non-breastfeeding women aged ≤ 35 years (at the time of trial enrollment).
  The PI calculation was based on the following formula:
  PI(evaluable cycles)= (∑ on-drug confirmed pregnancy ∈{exposure cycles})/(#{exposure cycles} ) X 1300
Time Frame: up to 13 months
Population: The population includes all non-breastfeeding subjects aged ≤ 35 years who were randomized, received at least one dose of study drug with sexual activity without using back-up contraception.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | Drospirenone 4 mg
Number analyzed (Participants) | 915
Pearl Index | 2.9 [1.5 to 5.1]

2. Secondary Outcome: Number of Pregnancies (All)
Description: Pearl Index based on overall cycles (overall PI) in women aged ≤ 35 years (at the time of trial enrollment) (confirmed pregnancies)
Time Frame: up to 13 months
Population: The population includes all non-breastfeeding subjects aged ≤ 35 years who were randomized and received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | LF111 (Drospirenone)
Number analyzed (Participants) | 915
Pearl Index | 2.7 [1.4 to 4.7]

3. Secondary Outcome: Number of Pregnancies (Method Failures)
Description: PI for method failures in women aged ≤ 35 years (at the time of trial enrollment) (confirmed pregnancies)
Time Frame: up to 13 months
Population: The population includes all non-breastfeeding subjects aged ≤ 35 years who were randomized, received at least one dose of study drug and used the IMP correctly.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | LF111 (Drospirenone)
Number analyzed (Participants) | 915
Pearl Index | 3.4 [1.4 to 7.0]

4. Secondary Outcome: Pregnancy Ratio
Description: Pregnancy ratio in women aged ≤ 35 years (at the time of trial enrollment)
Time Frame: up to 13 months
Population: The population includes all subjects aged ≤ 35 years who were randomized, received at least one dose of study drug with evaluable cycles.
Measure: Number (95% Confidence Interval); unit: Cumulative Pregnancy Rate (%)
Arm/Group | LF111 (Drospirenone)
Number analyzed (Participants) | 915
Cumulative Pregnancy Rate (%) | 2.46 [0.87 to 4.03]

5. Secondary Outcome: Overall PI, PI for Method Failures
Description: Overall PI, PI for method failures, PI (using evaluable cycles) and pregnancy ratio (life table analysis) in all women and in women up to 13 months (confirmed pregnancies)
Time Frame: up to 13 months
Population: The population includes all ages subjects who were randomized and received at least one dose of study drug, non-breastfeeding women and used the IMP correctly.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | LF111 (Drospirenone)
Number analyzed (Participants) | 993
Pearl Index | 2.9 [1.2 to 6.1]

6. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Description: Adverse events and changes in vital signs, clinical laboratory parameters
Time Frame: up to to 13 months
Population: The population includes all subjects who received at least one dose of the IMP.
Measure: Number; unit: Subjects
Arm/Group | LF111 (Drospirenone)
Number analyzed (Participants) | 1006
Subjects | 667

7. Secondary Outcome: Tolerability; Vaginal Bleeding Pattern
Description: Vaginal bleeding pattern
Time Frame: up to 13 months
Population: The population includes all subjects in full analysis set with bleeding.
Measure: Number; unit: Subjects with bleeding
Arm/Group | LF111 (Drospirenone)
Number analyzed (Participants) | 662
Subjects with bleeding | 505

8. Other Pre Specified Outcome: Number of Pregnancies (by BMI and Weight)
Description: PI for evaluable cycles in women aged ≤ 35 years in total and by BMI and weight subgroups based on confirmed and on confirmed and suspected, non-confirmed pregnancies
Time Frame: up to 13 months
Population: The population includes evaluable cycles in non-breastfeeding women aged ≤ 35 years , who were randomized and received at least one dose of study drug, including confirmed and suspected, non-confirmed pregnancies.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | LF111 (Drospirenone)
Number analyzed (Participants) | 915
Pearl Index
  Pearl Index BMI<30 | 4.1 [2.0 to 7.3]
  Pearl Index BMI>=30 | 2.9 [0.8 to 7.3]
  Weight < Median | 5.1 [2.4 to 9.3]
  Weight >= Median | 2.3 [0.8 to 5.5]

9. Other Pre Specified Outcome: Overall Pregnancies
Description: Overall PI based on confirmed and on confirmed and suspected, non-confirmed pregnancies in total and by BMI and weight subgroups
Time Frame: up to 13 months
Population: The population includes all ages subjects, non-breastfeeding women, who were randomized and received at least one dose of study drug, including confirmed and suspected, non-confirmed pregnancies.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | LF111 (Drospirenone)
Number analyzed (Participants) | 993
Pearl Index
  Pearl Index BMI<30 | 3.3 [1.7 to 6.0]
  Pearl Index BMI>=30 | 2.3 [0.6 to 5.8]
  Weight < Median | 4.2 [2.0 to 7.7]
  Weight >= Median | 1.9 [0.6 to 4.4]

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Drospirenone 4mg: Single treatment arm receives LF111 film-coated tablets (24 white tablets containing 4.0 mg drospirenone, 4 green placebo tablets), oral administration once daily.
Arm/Group | Drospirenone 4mg
All-Cause Mortality (participants affected / at risk) | 0/1006
Serious Adverse Events (participants affected / at risk) | 17/1006
Other Adverse Events (participants affected / at risk) | 341/1006
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drospirenone 4mg (N=1006)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 5
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1
DRUG ABUSE (Psychiatric disorders) | 1
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1
APPENDICITIS (Infections and infestations) | 1
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1
BILIARY COLIC (Hepatobiliary disorders) | 1
CELLULITIS (Infections and infestations) | 1
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1
INDUCED LABOUR (Pregnancy, puerperium and perinatal conditions) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Drospirenone 4mg (N=1006)
Metrorrhagia (Reproductive system and breast disorders) | 52
Dysmenorrhoea (Reproductive system and breast disorders) | 44
Breast pain (Reproductive system and breast disorders) | 43
Breast tenderness (Reproductive system and breast disorders) | 30
Menorrhagia (Reproductive system and breast disorders) | 17
Vaginal haemorrhage (Reproductive system and breast disorders) | 12
Amenorrhoea (Reproductive system and breast disorders) | 11
Menstruation irregular (Reproductive system and breast disorders) | 8
Vulvovaginal dryness (Reproductive system and breast disorders) | 5
Nausea (Gastrointestinal disorders) | 40
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal distension (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 7
Headache (Nervous system disorders) | 47
Migraine (Nervous system disorders) | 7
Acne (Skin and subcutaneous tissue disorders) | 30
Alopecia (Skin and subcutaneous tissue disorders) | 6
Weight increased (Investigations) | 23
Blood potassium increased (Investigations) | 5
Libido decreased (Psychiatric disorders) | 11
Mood swings (Psychiatric disorders) | 10
Depression (Psychiatric disorders) | 7
Affect lability (Psychiatric disorders) | 6
Irritability (Psychiatric disorders) | 5
Vulvovaginal mycotic infection (Infections and infestations) | 8
Fungal infection (Infections and infestations) | 5
Vulvovaginal candidiasis (Infections and infestations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 6
Hot flush (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT02269241/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT02269241/SAP_001.pdf